CLINICAL TRIAL: NCT02178657
Title: Intra-arterial Autologous Bone-marrow Mononuclear Cells Infusion for Acute Ischemic Stroke. A Phase II, Open-label, Multicenter, Randomized and Controlled Clinical Trial.
Brief Title: Intra-arterial Bone-marrow Mononuclear Cells Infusion for Acute Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andalusian Initiative for Advanced Therapies (Other Government)
Responsible Party: Principal Investigator, Francisco Moniche, Neurologist, Hospitales Universitarios Virgen del Rocío
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT 2013-002135-15; NCT02290483 (obsolete NCT alias)
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Cell therapy; Bone marrow
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bone marrow transplantation low dose (Experimental): Intra-arterial autologous bone marrow mononuclear cells injection (dose 2x10^6 per kilogram)
  Interventions: Drug: Autologous bone marrow mononuclear cell intra-arterial injection
- Bone marrow transplantation high dose (Experimental): Intra-arterial autologous bone marrow mononuclear cells injection (dose 5x10^6 per kilogram)
  Interventions: Drug: Autologous bone marrow mononuclear cell intra-arterial injection
- Control (No Intervention)

INTERVENTIONS:
Drug: Autologous bone marrow mononuclear cell intra-arterial injection
  Arms: Bone marrow transplantation high dose; Bone marrow transplantation low dose

SUMMARY:
This trial aims to test that intra-arterial injection of autologous bone marrow mononuclear cells in acute ischemic stroke patients is safe and improves neurological outcomes.

DETAILED DESCRIPTION:
This is a study in which the patients will be included diagnosed of ischemic stroke sharply in the territory of the cerebral average artery that there fulfill criteria of incorporation and none of those of exclusion and that they have signed the informed assent. 76 patients will randomize in proportion 2:1:1 in a group control that will receive only medical conventional treatment and in two groups of intervention that will receive an unique intra-arterial infusion of mononuclear autologous bone marrow stem cells (one group of dose of 2 millions of BMSC for kilogram of weight and another group of dose of 5 millions of BMSC for kilogram of weight). The three groups of patients will be followed for 24 months. The randomization will be stratified depending on the NHSS score. This clinical trial has a voluntary substudy to obtain information on plasma biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with middle cerebral artery (MCA) acute ischemic stroke.
* Time of stroke onset is known and treatment can be started between day 1 and 7 of onset.
* DWI-MRI has reliably shown acute MCA ischemic lesions
* Magnetic resonance angiography (MRA) must confirm ipsilateral MCA permeability
* National Institute of Health Stroke Scale score of 6-20 at inclusion
* Age 18-80 years
* Written informed consent has been obtained

Exclusion Criteria:

* Hemorrhagic stroke or symptomatic hemorrhagic transformation
* Lacunar infarction
* Preocclusive stenosis or total occlusion of ipsilateral carotid artery
* Worsening of ≥4 points in National Institute of Health Stroke Scale in the 24 hours previous to inclusion, attributable to edema or hemorrhagic transformation or suspicious of malignant edema
* Decrease of consciousness with a Glasgow Coma Scale of <8 points
* Patients with present or previous malignant disease during the last 5 years, except for basal cell carcinoma
* Contraindication for MRI or for bone marrow harvest
* Previous diagnosis of neurodegenerative disease
* Acute heart failure
* Hepatic or renal dysfunction (creatinine >2mg/dL)
* Coagulopathy
* Severe co-morbidity
* Pregnancy, childbearing potential (unless it is certain that pregnancy is not possible) or breast feeding
* Modified Rankin Score (mRS) before stroke of ≥2
* Participation in any clinical trial in the last 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-04; Primary Completion 2021-10-27 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Disability | 6 months
  Proportion of patients with modified Rankin Scale scores of 0-2 at 6 months

SECONDARY OUTCOMES:
Mortality | 24 months

OTHER OUTCOMES:
Functional outcomes | 6 months
  Functional outcome measure by National Institute of Health Stroke Scale and Barthel at 6 months
Infarct volume | 6 months
  Infarct volume change between baseline (DWI) and 6 months (FLAIR)
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 24 months
Number of Participants with new-onset seizures as a Measure of Safety and Tolerability | 6 months
Functional outcomes | 6 months
  Categorical shift in mRS ordinal (0-6) scale

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Moniche, MD, PhD, Principal Investigator — Hospitales Universitarios Virgen del Rocio
Locations (4):
- Spain (4):
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospitales Universitarios Virgen del Rocio, Seville
  - Hospitales Universitarios Virgen Macarena, Seville

REFERENCES:
- [Derived] Cabezas-Rodriguez JA, Biarnes C, Marti-Navas M, Pineda V, Comas-Cufi M, Pardo-Galiana B, Zapata-Arriaza E, Pinero P, Aguera-Morales E, Valverde R, Ortega-Quintanilla J, Ainz-Gomez L, Baena-Palomino P, Gutierrez I, Medina-Rodriguez M, Ocete-Perez R, Gamero MA, de Alboniga-Chindurza A, Hermosin A, Aguilar-Perez M, Villagran D, Escamilla-Gomez V, Calderon-Cabrera C, Nogueras S, Jimenez R, Martin V, Herrera C, Delgado F, Gonzalez A, Montaner J, Puig J, Moniche F. Diffusion Tensor Imaging Study After Intraarterial Cell Therapy in Acute Ischemic Stroke: A Substudy of the IBIS Randomized Clinical Trial. Stroke. 2025 Aug;56(8):2198-2209. doi: 10.1161/STROKEAHA.124.050261. Epub 2025 Apr 30. PMID 40304033
- [Derived] Moniche F, Cabezas-Rodriguez JA, Valverde R, Escudero-Martinez I, Lebrato-Hernandez L, Pardo-Galiana B, Ainz L, Medina-Rodriguez M, de la Torre J, Escamilla-Gomez V, Ortega-Quintanilla J, Zapata-Arriaza E, de Alboniga-Chindurza A, Mancha F, Gamero MA, Perez S, Espinosa-Rosso R, Forero-Diaz L, Moya M, Pinero P, Calderon-Cabrera C, Nogueras S, Jimenez R, Martin V, Delgado F, Ochoa-Sepulveda JJ, Quijano B, Mata R, Santos-Gonzalez M, Carmona-Sanchez G, Herrera C, Gonzalez A, Montaner J. Safety and efficacy of intra-arterial bone marrow mononuclear cell transplantation in patients with acute ischaemic stroke in Spain (IBIS trial): a phase 2, randomised, open-label, standard-of-care controlled, multicentre trial. Lancet Neurol. 2023 Feb;22(2):137-146. doi: 10.1016/S1474-4422(22)00526-9. PMID 36681446
- [Derived] Mancha F, Escudero-Martinez I, Zapata-Arriaza E, Vega-Salvatierra A, Cabezas JA, Lebrato L, Pardo B, De-La-Torre J, Zapata M, Escamilla V, Calderon-Cabrera C, Martin-Sanchez J, Valverde R, Aguera-Morales E, Herrera I, Delgado F, Gamero MA, Perez-Sanchez S, Moya M, Espinosa R, Ortega-Quintanilla J, Gutierrez-Jarrin I, Gonzalez-Garcia A, Montaner J, Moniche F. Circulating microRNA after autologous bone marrow mononuclear cell (BM-MNC) injection in patients with ischemic stroke. J Investig Med. 2020 Mar;68(3):807-810. doi: 10.1136/jim-2019-001161. Epub 2019 Dec 17. PMID 31852749
- [Derived] Moniche F, Escudero I, Zapata-Arriaza E, Usero-Ruiz M, Prieto-Leon M, de la Torre J, Gamero MA, Tamayo JA, Ochoa-Sepulveda JJ, Maestre J, Carmona M, Pinero P, Calderon-Cabrera C, Jimenez MD, Gonzalez A, Montaner J. Intra-arterial bone marrow mononuclear cells (BM-MNCs) transplantation in acute ischemic stroke (IBIS trial): protocol of a phase II, randomized, dose-finding, controlled multicenter trial. Int J Stroke. 2015 Oct;10(7):1149-52. doi: 10.1111/ijs.12520. Epub 2015 Jun 4. PMID 26044701